CLINICAL TRIAL: NCT00800098
Title: Effects of an Herbal Topical Cream on Osteoarthritis Symptoms, Biomarkers, and Disease Progression in the Knee
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anne Friedlander, Consulting Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SU-11252008-1355; Protocol ID:14764
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo cream matched on consistency, color, and smell
  Interventions: Drug: herbal topical cream
- Active (Active Comparator): AARP active arthritis cream
  Interventions: Drug: herbal topical cream

INTERVENTIONS:
Drug: herbal topical cream

SUMMARY:
Arthritis Relief Plus (ARP) Cream is a natural, herbal cream that has been shown to provide pain relief and decreased stiffness. Anecdotal reports suggest that pain may continue to be reduced months after cream use is stopped, indicating that there could be some disease-modifying effects of the cream. The purpose of this study is to test the claim that the ARP cream can provide long-term pain relief to osteoarthritis patients after only a short period of use. The study will also try to determine whether the pain relief is accompanied with any measurable indications that the progression of osteoarthritis has slowed or halted

DETAILED DESCRIPTION:
General Procedure: Subjects will be screened for: a history of knee pain and surgery by questionnaire; kidney disease as determined by blood creatinine levels; knee diameter less than 17cm and body diameter less than 60 cm due to the physical constraints of the MRI. Prior X-rays or MRIs will be examined to evaluate the subject's level of OA. X-rays and MRIs that are older than 2 years, cannot be used and these potential subjects will receive one set of 2 knee x-rays prior to enrollment. If they qualify and wish to enroll, they will be matched on age, sex and degree of OA and assigned by a 3rd party investigator to either a placebo group or active treatment group. Subjects will be asked to complete baseline questionnaires, functional tests, and have blood draws and MRI screenings before starting their treatment. Enrolled subjects will apply 2.5 grams of active or placebo cream 3 times per day to the skin over the affected knee for 12 weeks. Further measurements will be taken periodically throughout the course of the study, as detailed below.

MRI: Subjects will receive MRI scans of the affected knee 3 times: at enrollment, 12 weeks, and 15 months. The MRI scan sessions will take place at the Lucas Center for MRI at Stanford University. In preparation for the MRI scan, subjects will be required to fill out a standard MRI screening form to ensure that there are no conditions that could interfere with the MRI imaging or that could make scanning in any way hazardous. During the sessions, subjects will lie on the scanner table on their backs with their legs straight. We will scan one knee. The time for this scan will be approximately 1 hour. This entire session will take approximately 1 and 1/2 hours, including setup time.

Subjects may be asked to receive a small dose of intravenous gadolinium contrast agent, administered by Dr. Gold. This is to improve the evaluation of the articular cartilage.

Questionnaires: Subjects will receive physical activity, pain and function questionnaires at enrollment, 4 weeks, 8 weeks, 12 weeks, 14 weeks, 16 weeks, 20 weeks, 6 months, 9 months, 12 months, and 15 months. They will also keep a log of use of other pain medicine, such as aspirin.

Blood/Urine Samples: A small amount of blood (2 tablespoons or 30 ml) will be drawn and urine collected up to 11 times throughout the investigation to study blood markers of cartilage breakdown (COMP, CTX2, Glc-Gal-PYD) and synthesis (PIIANP) as well as inflammation (HA, CRP) and joint vascularity (TNF-alpha, IL-6, osteocalcin). Blood creatinine levels will be tested at baseline only.

Functional Testing: Subjects will also participate in functional testing that will include walking tests, rising from a chair, and climbing stairs up to 11 times throughout the 15-month study. The "6-minute Walk" test is a good indicator of cardiovascular capacity. We will ask subjects to cover as much ground as possible in 6 minutes at a maintainable pace, and will record the distance traveled. The "Get up and Go" test will measure the time it takes a subject to rise from a standard chair, walk three meters, turn around, return, and sit down again. Subjects will perform 3 trials, and their fastest time will be recorded. The "Timed Stair Climb" test will measure the time it takes subjects to climb up and down five standardized steps. Subjects will be instructed to ascend and descent as fast as possible using the handrails provided. They will perform 3 trials and the fastest time will be selected. Walking speed tests offers an indirect way to measure the functional impact of pain. We will ask subjects to walk 10 meters at a maximal or a self-selected pace and will calculate their walking speeds. They will perform between 3 to 6 trials of each test.

All tests will be performed in accordance with ACSM guidelines for exercise testing.

ELIGIBILITY:
Inclusion Criteria:-Men and women between 40-70 years old

* Have a history of knee pain
* Exhibit mild osteoarthritis on the knee, as determined by Dr. Gold through MRIs and radiographs (if available). Exclusion Criteria:-Outside of age range
* Prior knee surgery
* History of knee or knee ligament instability
* History of intermittent or persistent knee joint swelling
* History of trauma to the knee or lower extremities resulting in fracture, tears of menisci, ligaments or joint capsule, or cartilage damage
* Unable to have MRI scan due to the presence of metallic internal devices that would represent a risk factor for MRI and known or suspected pregnancy.

History of corticosteroid use

* Kidney Disease
* Knee diameter greater than 17cm and body diameter greater than 60 cm due to the physical constraints of the MRI

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
WOMAC | 12 weeks

SECONDARY OUTCOMES:
Function | 12 weeks
MRI morphology | 12 weeks
Blood and urine biomarkers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne L. Friedlander, Principal Investigator — Stanford University; Garry Evan Gold, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States